CLINICAL TRIAL: NCT06816784
Title: COMPARISON OF OUTCOME OF AUTOLOGOUS SERUM THERAPY VS LEVOCETRIZINE IN THE TREATMENT OF CHRONIC URTICARIA
Brief Title: Treatment Options for Chronic Urticaria
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Sheikh Zayed Medical College (Other Government)
Responsible Party: Principal Investigator, Farah Humera, post graduate resident indermatology, Sheikh Zayed Medical College
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: sheikh-ZMCFH
Record Dates: First submitted 2025-01-21; First posted 2025-02-10 (Actual); Last update posted 2025-02-10 (Actual); Status verified 2025-02

CONDITIONS: Chronic Urticaria
Keywords: chronic urticaria; autologous serum therapy; levocetrizine
MeSH Terms: conditions — Chronic Urticaria | interventions — levocetirizine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Autologous serum therapy group (Active Comparator): Group A will receive AST 5 ml of blood will be collected and centrifuged at 3000 r.p.m for 10 min to obtain serum,2 ml of the serum will be injected into the gluteus muscle. We will give the patients injection of Autologous Serum intramuscularly once a week for 9weeks
  Interventions: Drug: Autologous serum therapy
- levocetirizine group (Active Comparator): Group B will receive levocetirizine orally 5mg one tablet HS
  Interventions: Drug: Oral levocetirizine

INTERVENTIONS:
Drug: Autologous serum therapy — 5 ml of blood will be collected and centrifuged at 3000 r.p.m for 10 min to obtain serum,2 ml of the serum will be injected into the gluteus muscle. We will give the patients 9 injections of Autologous Serum intramuscularly once a week
  Arms: Autologous serum therapy group
Drug: Oral levocetirizine — Group B will receive oral levocetirizine 5mg 1 tablet HS.
  Arms: levocetirizine group

SUMMARY:
chronic urticaria is one of the most common dermatological disease affecting many people, exploring most treatment options for its treatment is need of an hour.

Our study aim to compare the efficacy of Autologous Serum Therapy (AST) with levocetirizine in Chronic Urticaria patients

DETAILED DESCRIPTION:
Urticaria is one of the most common skin diseases causing redness, and swelling in the dermis and epidermal layers and are severely pruritic.

Chronic urticaria is further sub-divided into chronic spontaneous urticaria and chronic inducible urticaria. International guidelines recommend non-sedating antihistamines once daily as first-line therapy for chronic spontaneous urticaria and chronic inducible urticaria.

Levocetirizine which is classified as a second-generation antihistamine and works by blocking histamine H1-receptors , is an effective treatment for CIU, characterized not only by a rapid and sustained response, but also by an important improvement in QOL.

Autologous serum therapy (AST) has been tried by many in patients with CAU with variable results, majority showing beneficial effects. AST has also been used in the treatment of ocular alkali burn patients Presence of tolerance generating anti-idiotype antibodies to mast cell degranulating antigens that induce remission of the disease forms the basis of AST and this therapy has been tried in various autoimmune diseases Our study aim to compare the efficacy of Autologous Serum Therapy (AST) with levocetirizine in Chronic Urticaria patients OBJECTIVE "TO COMPARE THE EFFICACY OF AUTOLOGOUS SERUM THERAPY VS LEVOCETRIZINE IN THE TREATMENT OF CHRONIC URTICARIA IN TERTIARY CARE HOSPITAL"

DATA COLLECTION:

Data will be collected on prescribed proforma which is attached, at Dermatology OPD, Sheikh Zayed Hospital, Rahim Yar Khan. Patient will be selected on basis of inclusion & exclusion criteria. Informed consent will be taken from selected patients before data collection. Study will include 72 patients which will be divided into 2 groups, A & B, 36 in each group. Group A will receive AST, Group B will receive oral levocetirizine 5mg 1 tablet HS.

5 ml of blood will be collected and centrifuged at 3000 RPM for 10 min to obtain serum,2 ml of the serum will be injected into the gluteus muscle. We will give the patients 9 injections of Autologous Serum intramuscularly once a week .

Follow up visit will be after 2 months of last session.

DATA ANALYSIS:

Data will be analyzed by SPSS v25.0

ELIGIBILITY:
Inclusion Criteria:

* Age: 13-60 years
* Gender: Both male and female
* Patients having urticaria for more than 6 weeks diagnosed clinically

Exclusion Criteria:

* Pregnancy and lactating females
* Patients who are immunosuppressed either due to medication or disease.
* Patients suffering from chronic diseases i-e chronic liver disease, chronic kidney disease.
* Patients taking steroids in last 2 weeks.

Ages: 13 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 72 (Estimated)
Dates: Start 2025-02 (Estimated); Primary Completion 2025-07 (Estimated); Study Completion 2025-07 (Estimated)

PRIMARY OUTCOMES:
COMPARISON OF OUTCOME OF AUTOLOGOUS SERUM THERAPY VS LEVOCETRIZINE IN THE TREATMENT OF CHRONIC URTICARIA | Clinical assessment for efficacy will be done monthly for 6 months
  Efficacy will be assessed clinically at each follow up visit. Final efficacy of each treatment will be determined at last follow up visit( i.e. at 7th week after start of treatment).The final efficacy will be divided into following groups on the basis of clinical resolution of disease: 1. Excellent efficacy: It is defined as greater than 80% reduction in the frequency of urticaria episodes per week as measured from baseline 2. moderate efficacy: It is defined as 50% to less than 80% reduction in number of urticaria episodes per week as measured from baseline healing of urticaria from the baseline. 3.non-efficaceos: It is defined as less than a 50% reduction in the frequency of urticaria episodes per week from baseline.

CONTACTS AND LOCATIONS:
Locations (1):
- Sheikh zayed Medical College and Hospital, Rahim Yar Khan, Punjab 644200, Rahim Yar Khan, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No